CLINICAL TRIAL: NCT03255863
Title: Determinants of Patients' Uptake of Therapeutic Education Programme
Acronym: UTEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2015_70; 2016-A02057-44 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2017-08-16; First posted 2017-08-21 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2020-08

CONDITIONS: Chronic Disease; Patient Education as Topic; Patient Adherence; Empathy; Quality of Healthcare
Keywords: Psychological Theory
MeSH Terms: conditions — Chronic Disease; Patient Compliance | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Questionnaire (Other): Auto and hetero questionnaire
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Patient Self reported questionnaire filled in.

SUMMARY:
Therapeutic Patient Education (TPE) refers to programs that help patients to manage life with a chronic disease in the best possible way. In spite of the effectiveness of Therapeutic Patient Education, few patients uptake TPE when it is proposed to them. Therefore, our main aim was to identify patients' beliefs that will predict patients' uptake of TPE. According to the Health Belief Model, patient will participate in TPE if they perceive their disease as a serious threat (with possible serious complications), but which can be controlled however, and that TPE is efficient and represents little burden.

Secondary aims are as follows:

1. To test whether the way TPE is presented to patients impact patients' decision to uptake TPE. The way TPE is presented comprises the time between diagnosis and the proposal of TPE, whether patient is a remission or crisis period in the disease, the time between the proposal and the next TPE session, and what is said by healthcare professionals to present TPE.
2. To test whether healthcare professionals' empathy impact patients' decision to participate in TPE
3. To test whether patients' intention to participate in TPE will predict their actual participation.

The ultimate goal of the study is to identify patients whose beliefs will not favor participation in TPE in order to accompany those patients more carefully. Best practices will be proposed according the results.

ELIGIBILITY:
Inclusion Criteria:

* Patients to whom TPE was proposed in diabetes, hemophilia, obesity, cardiac failure, chronic inflammatory bowel disease, parkinson, rare diseases, epilepsy, peripheral arterial diseases
* Belong to a social security scheme
* Pregnant women to whom TPE for gestational diabetes is proposed

Exclusion Criteria:

* Cognitive impairment declared by healthcare professionals
* Inpatients
* Patients for whom TPE is coupled with rehabilitation
* Psychiatric disorders
* Patients who cannot give informed consent
* Patients in jail

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 459 (Actual)
Dates: Start 2017-12-20 (Actual); Primary Completion 2020-09-09 (Actual); Study Completion 2020-09-09 (Actual)

PRIMARY OUTCOMES:
Patient's intention to participated in TPE by a questionnaire based on the Health Belief Model | Baseline (after TPE proposal)
  Patient's participation in TPE : yes or no Participation is defined as the patient's intention to come expressly to the hospital for a first appointment dedicated to therapeutic education.
  The main variables of the HBM will be analyzed: perceived threat of the pathology, perceived benefits and barriers to TPE, perceived patient control of its pathology.

SECONDARY OUTCOMES:
Time limit of first proposition in TPE | Baseline
  Time between date of diagnostic illness and date of first first proposition in TPE
Timeout of first participation in TPE | Baseline
  Time between date of proposition and date of the program begin of TPE
Medical context in which TPE is proposed | Baseline
  Medical context in acute phase versus phase of stabilization of the pathology
Consultation And Relational Empathy (CARE) questionnaire | Baseline
  The patient's perceived empathy of the professional (s) who offered the TPE will be assessed by the CARE questionnaire
Visual analog scale for intention to participated | Baseline
  Visual analog scale ranging from 0 "not at all intending to participate" to 100 "very strong intention to participate Measurement of the patient's intention to participate in the proposed TPE program

CONTACTS AND LOCATIONS:
Overall Officials: Maryline Bourgoin, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Claude Huriez, CHU, Lille, France

IPD SHARING:
Plan to Share IPD: No